CLINICAL TRIAL: NCT03887819
Title: The Dating of Thrombus Organization in Cases of Pulmonary Embolism: an Autopsy Study
Brief Title: Pulmonary Embolism: an Autopsy Study
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, clinical professor, University of Campania Luigi Vanvitelli
Other Study IDs: SecondUNI 21.03.2019
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — human tissue samples and pulmonary thrombi.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hystological evaluation — The original tissues samples will be fixed in 10% neutral buffered formalin and embedded in paraffin blocks. Sections (4 μm thick) will be stained with hematoxylin and eosin stain (H&E) for diagnosis. The immunohistochemistry for anti-LCA, anti-CD68, and anti-CD3 will be performed to identify the inflammatory infiltrate.

SUMMARY:
BACKGROUND: Pulmonary embolism (PE) is associated to high mortality rate worldwide. However, the diagnosis of PE often results inaccurate. Many cases of PE are incorrectly diagnosed or missed and they are often associated to sudden unexpected death (SUD). In forensic practice, it is important to establish the time of thrombus formation in order to determine the precise moment of death. The autopsy remains the gold standard method for the identification of death cause allowing the determination of discrepancies between clinical and autopsy diagnoses. The aim of our study will be to verify the morphological and histological criteria of fatal cases of PE and evaluate the dating of thrombus formation considering 5 ranges of time.

METHODS: Pulmonary vessels sections will be collected from January 2010 to December 2017. Sections of thrombus sampling will be stained with hematoxylin and eosin. The content of infiltrated cells, fibroblasts and collagen fibers will be scored using a semi-quantitative three-point scale of range values.

Hypothesis: After a macroscopic observation and a good sampling traditional histology, it will be important to identify the time of thrombus formation. We will identify histologically a range of time in the physiopathology of the thrombus (early, recent, recent-medium, medium, old), allowing to determine the dating of thrombus formation and the exact time of death.

DETAILED DESCRIPTION:
Introduction Venous thromboembolism (VTE) is pathological condition caused by deep vein thrombosis (DVT) with a consequent detaching of thrombus from original sites , that by embolic phenomena and traveling to the lung might result in pulmonary embolism (PE). As first, the diagnosis of PE might result frequently inaccurate, with many cases incorrectly diagnosed or missed. Secondly, it might be caused by several conditions such as surgery and trauma, with a consequent relevant clinical impact and worse prognosis. However, clinical presentation of PE range from those completely asymptomatic or with an insidious disease, to sudden unexpected death (SUD. SUD may be defined as a natural and fatal event that occurs within 1 h of the beginning of symptoms in an apparently healthy subject or in those with a disease not particularly severe to cause an abrupt outcome. Since the diagnosis is challenging, epidemiological data regarding PE mortality remain limited.To date, it is estimated that PE is responsible for 100,000 annual deaths only in the United States and approximately 25-30% of patients had SUD as consequence of PE.

However, in our opinion it might be essential to collect morphological macroscopic evaluation elements to distinguish a thrombus from an embolus or agonic coagulum.To date, the autopsy may be useful for the determination of the identification of death cause, and to establish the dating of transformation of thrombus and evaluate any professional error. Therefore, in this study, authors will critically review the histological section of thrombus from 30 fatal cases of PE pulmonary embolus by autopsies, and its correlation and origin prior or subsequent to a traumatic event, as confirmed by post-mortem examination and final diagnosis. Moreover, the aim of this study will be to evaluate the chronological transformation of the thrombus and to establish the time of death for each subject.

Materials and methods Patients and samples Pulmonary vessels sections will be collected from 30 fatal cases of PE (25 cases of hospitalized patients and 5 cases of SUD) defined according to commonly accepted criteria were routinely collected from January 2010 to December 2017 at the University of Naples Federico II.

Histological evaluation According to the guidelines for autopsy from the Association for European Cardiovascular Pathology, and in all cases authors will examine the pulmonary arterial trunk by posterior approach. Sections (4 μm thick) will be stained with hematoxylin and eosin stain (H&E) for diagnosis. The original tissues samples will be fixed in 10% neutral buffered formalin and embedded in paraffin. The immunohistochemistry for anti-LCA, anti-CD68, and anti-CD3 will be performed to identify the inflammatory infiltrate. In addition, authors will be performed an immunofluorescence method to identifying the deposition of factor VIII and fibrinogen. A Picro Sirius Red/Fast Green will be used for differential staining of collagen during matrix production phase. All stained samples will be examined under infiltrate, absent or rare lympho-monocytic inflammatory elements. The vessels of small and medium will be involved, mainly from the main branches of the pulmonary vessels.In2 patients we observed a score 3 for cellular infiltrate and 1 for fibrosis. In 10 cases (5 heart patients, 2 cardiac patients undergoing surgery and 3 surgeries), authors will observe an increase (score 2) in the digital and light microscope.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute pulmonary embolism;
* patients died after the pulmonary embolic event.

Exclusion Criteria:

* diagnosis of non acute pulmonary embolism;
* patients survived after the pulmonary embolic event.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include 19 male (63.3%) and 11 female (36.7%). Their age will range from 38 to 87 years.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
To evaluate pulmonary thrombus burden | 24 months
  Authors will evaluate if a pulmonary embolus was originated prior or subsequent to a traumatic event. However, they will evaluate the dimension of the thrombus, and the quantity of fibrinogen present in the thrombus, from pulmonary vessels sections. The tissues samples will be fixed in 10% neutral buffered formalin and embedded in paraffin blocks, and stained with hematoxylin and eosin stain for diagnosis. For inflammatory cellular infiltration and fibrosis, authors will attribute a score 0 for no increase, score 1, 2, or 3 for little, moderate, or high increase of cell content compared to adjacent tissue, respectively. For the extracellular matrix production, authors will attribute a score 0 for absence of collagen production, score 1 and 2 for 10-40% and 40-80% collagen fibers content compared to adjacent normal tissue, respectively, and finally score 3 for wound matrix indistinguishable from adjacent normal tissue.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mansueto G, Costa D, Capasso E, Varavallo F, Brunitto G, Caserta R, Esposito S, Niola M, Sardu C, Marfella R, Napoli C, Paternoster M. The dating of thrombus organization in cases of pulmonary embolism: an autopsy study. BMC Cardiovasc Disord. 2019 Nov 8;19(1):250. doi: 10.1186/s12872-019-1219-8. PMID 31703628